CLINICAL TRIAL: NCT01751412
Title: Pilot Study Evaluating the Use of Proton Radiation for Treatment of Lymphoma Involving the Mediastinum
Brief Title: Proton Radiation for Lymphoma Involving Mediastinum
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow accrual rates/ lack of funding
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Tom DeLaney, MD, Medical Director, Francis H. Burr Proton Therapy Center, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-346
Record Dates: First submitted 2012-12-14; First posted 2012-12-18 (Estimated); Results first posted 2017-10-17 (Actual); Last update posted 2017-11-24 (Actual); Status verified 2017-10

CONDITIONS: Lymphoma
Keywords: Hodgkin; Non-Hodgkin Lymphoma; Mediastinal; Adult Lymphoma; Pediatric Lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Non-Hodgkin | interventions — Proton Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Proton Radiation (Experimental): Delivered daily (Monday-Friday) for two to five weeks.
  Interventions: Radiation: Proton Radiation

INTERVENTIONS:
Radiation: Proton Radiation

SUMMARY:
This research study is a Pilot Study. Pilot studies are conducted to see if it is practical to do this type of research on a larger scale in the future. The pilot part of this study is to assess the possibility of using proton radiation to treat lymphomas. Proton radiation is used for many other types of malignancies, but its use for the treatment of lymphoma has been limited. The treatment is still being studied as research doctors are trying to find out more about its use in the treatment of different types of lymphoma. Proton beam radiation therapy is an FDA approved radiation delivery system.

Patients are being asked to participate in this research study if they have lymphoma in the center of their chest, near their heart. Conventional radiation therapy with photons is used as standard treatment for many patients with lymphoma. In this research study investigators are looking at another type of radiation called proton radiation, which is known to spare surrounding tissue and organs from radiation. Proton radiation delivers radiation to the area requiring radiation but delivers no dose beyond the region requiring treatment. This may reduce side effects that patients would normally experience with conventional radiation therapy or other means of delivering proton radiation therapy.

In this research study, investigators are evaluating the effectiveness of using proton radiation delivered to reduce side effects associated with radiation treatment.

DETAILED DESCRIPTION:
If a person agrees to participate in this research study, they will be asked to undergo some screening tests or procedures to confirm eligibility. Many of these tests and procedures are likely to be part of regular cancer care and may be done even if it turns out that a patient does not take part in the research study. If a patient has had some of these tests or procedures recently, they may or may not have to be repeated. These tests and procedures include: a medical history, performance status, physical examination, assessment of tumor, echocardiogram, electrocardiogram, pulmonary (lung) function tests and blood tests. If these tests show that a patient is eligible to participate in the research study, they will begin the study treatment. If a patient does not meet the eligibility criteria, they will not be able to participate in the research study.

Proton radiation will be delivered daily for 2 to 5 weeks, depending on the dose prescribed by your physician. Treatment is delivered (Monday-Friday) for 5 days (no weekends or holidays). Each treatment will require that you lie on a table for 30 to 45 minutes.

Participants will receive radiation therapy as an outpatient at Massachusetts General Hospital. During radiation therapy, they will have the following weekly assessments and procedures: physical exam, assess for any side effects, blood tests for cardiac markers.

Study participants will be asked to return for a follow up visit 6-12 weeks after their last dose of radiation therapy. During this visit the following tests and procedures will be done: PET/CT scan, physical exam, assess for side effects and blood tests for cardiac markers.

Participants will also be asked to return for a follow-up visit at 6 months, 12 months and annually for five years post radiation. Keeping in touch with study participants and checking on their condition helps investigators look at the long-term effects of the research study. At these visits, the following tests and procedures will be done: physical exam, assess for any side effects, ECG, ECHO, pulmonary tests, PET/CT scan, routine blood tests and blood tests for cardiac markers (at 6 months and 1 years only).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed Hodgkin lymphoma or non-Hodgkin lymphoma
* Must complete standard chemotherapy appropriate for the histologic subtype of lymphoma and be able to start radiation therapy within 3-6 weeks of completing chemotherapy
* Life expectancy of at least 12 months
* Must have achieved complete or partial response per appropriate imaging technique within 4 weeks of study entry following administration of chemotherapy
* Individuals with known history of HIV positivity must be on appropriate HAART therapy

Exclusion Criteria:

* Pregnant or breastfeeding
* Prior therapeutic radiation therapy > 200 cGy has been delivered to target volume
* Have not recovered from adverse events due to systemic agents administered more than 4 weeks earlier
* Uncontrolled intercurrent illness
* History of a different malignancy unless disease free for at least 2 years (cervical cancer in situ, basal or squamous cell carcinoma are acceptable)
* Receiving any other investigational agents

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas DeLaney, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Proton Radiation: Proton Radiation, delivered daily (Monday-Friday) for two to five weeks.
Period: Overall Study
Arm/Group | Proton Radiation
Started | 12
Completed | 11
Not Completed | 1
Not completed — Disease Progression Before Treatment | 1

BASELINE CHARACTERISTICS:
Arm/Group | Proton Radiation
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 11
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 28 [17 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Mean Radiation Dose to Normal Heart Tissue
Description: The mean radiation dose to the heart in Gy RBE (Gray relative biological effectiveness).
Time Frame: 6 weeks
Measure: Mean (Full Range); unit: Gy(RBE)
Arm/Group | Proton Radiation
Number analyzed (Participants) | 12
Gy(RBE) | 5.4 [1.63 to 17.13]

2. Primary Outcome: Radiation Dose to the Normal Tissue of the Lungs
Description: The percentage of the lung volume which received radiation dose of 20 Gray (Gy) or more. The lung volume percentages for the 12 participants were averaged and presented separately for the left and right lungs.
Time Frame: 6 Weeks
Measure: Mean (Full Range); unit: Percentage of Lung Volume
Arm/Group | Proton Radiation
Number analyzed (Participants) | 12
Percentage of Lung Volume
  Left Lung | 9.17 [3.27 to 20.22]
  Right Lung | 8.79 [2.38 to 16.48]

3. Secondary Outcome: Local Control
Description: The number of participants who maintained local control for the duration of their followup. Local control is defined as the lack of disease progression. Progression is the increased growth of cancer cells or the spread of the cancer cells to another location within the body.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Proton Radiation
Number analyzed (Participants) | 12
Participants | 10

4. Secondary Outcome: Number of Participants With Acute Toxicities
Description: Acute toxicities including pericarditis, pneumonitis, Lhermitte's, dermatitis, mucositis, esophagitis, leukopenia, xerostomia, and thrombocytopenia. Data is shown as the number of participants that experienced the given toxicities.
Time Frame: 90 Days
Measure: Number; unit: participants
Arm/Group | Proton Radiation
Number analyzed (Participants) | 12
participants
  pericarditis | 0
  pneumonitis | 0
  Lhermitte's | 0
  dermatitis | 9
  mucositis | 0
  esophagitis | 2
  leukopenia | 0
  xerostomia | 0
  thrombocytopenia | 0

5. Secondary Outcome: Late Toxicities
Description: Late toxicities including clinical and sub-clinical heart disease, pulmonary fibrosis, esophageal stricture, myelopathy, thyroid dysfunction and secondary cancers.
Time Frame: 5 years
Population: The trial was terminated before the study endpoint was met. The data is not available for analysis.
Arm/Group | Proton Radiation
Number analyzed (Participants) | 0

6. Secondary Outcome: 6-Month Overall Survival
Description: The number of participants surviving six months after starting treatment
Time Frame: 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Proton Radiation
Number analyzed (Participants) | 12
Participants | 12

7. Secondary Outcome: 6-Month Progression-Free Survival
Description: The number of participants surviving without disease progression six months after the start of treatment
Time Frame: 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Proton Radiation
Number analyzed (Participants) | 12
Participants | 12

ADVERSE EVENTS:
Time Frame: Weekly during radiation therapy. After completion of therapy at 6-12 weeks , 6 months, and annually during follow-up. Patients are followed for 5 years or until death, whichever occurs first. Study was terminated before planned and participants were only followed for a median duration of 2 years.
Description: Toxicity is evaluated with physical exams; cardiology exams (Echocardiogram and Electrocardiogram); pulmonary function tests (Diffusing capacity of the lungs for carbon monoxide (DLCO), forced exhaled volume in 1 second (FEV 1) and FEV1 / FVC (forced vital capacity); and laboratory tests.
Arm/Group | Proton Radiation
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 9/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Proton Radiation (N=11)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 3 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dermatitis radiation (Injury, poisoning and procedural complications) | 9 (10)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Esophageal obstruction (Gastrointestinal disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 6 (8)
Forced expiratory volume decreased (Investigations) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3 (3)
General disorders and administration site conditions - Other, specify (General disorders) | 2 (2)
Headache (Nervous system disorders) | 1 (1)
Hot flashes (Vascular disorders) | 2 (2)
Hypertension (Vascular disorders) | 1 (1)
Immune system disorders - Other, specify (Immune system disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Irregular menstruation (Reproductive system and breast disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain (General disorders) | 2 (2)
Palpitations (Cardiac disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Thromboembolic event (Vascular disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Weight loss (Investigations) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated prematurely due to funding issues. Limited enrollment and shorter than planned follow-up prevented statistically significant evaluation of endpoints.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes